CLINICAL TRIAL: NCT00141791
Title: A Randomized, Double-Blind, Placebo Controlled Trial Evaluating the Safety and Efficacy of Etanercept 25mg Twice Weekly in Subjects With Moderate to Severe Persistent Asthma
Brief Title: Study Evaluating Etanercept in Moderate to Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A8-205
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Asthma
Keywords: Asthma; Anti-Asthmatic Agents; Receptors; Tumor Necrosis Factor
MeSH Terms: conditions — Asthma | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The primary objective of the study is to assess the efficacy and safety of etanercept 25 mg given twice weekly in subjects with moderate to severe persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe persistent asthma for at least 1 year
* Demonstrated reversibility of at least 9% and (FEV1) 50% to 80% predicted
* Subjects must be on a high-dose inhaled corticosteroid (ICS)

Exclusion Criteria:

* Previous treatment with etanercept
* Current use of cigarettes
* Significant concurrent medical conditions at the time of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change in FEV1% predicted from baseline to week 12 (before bronchodilator administration).

SECONDARY OUTCOMES:
Peak expiratory flow rate, Asthma control questionnaire, Asthma exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (13):
- United States (13):
  - Birmingham, Alabama
  - Denver, Colorado
  - Sarasota, Florida
  - Tallahassee, Florida
  - Valrico, Florida
  - Covington, Louisiana
  - Wheaton, Maryland
  - Boston, Massachusetts
  - Rockville Centre, New York
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Richmond, Virginia
  - Madison, Wisconsin

REFERENCES:
- [Derived] Holgate ST, Noonan M, Chanez P, Busse W, Dupont L, Pavord I, Hakulinen A, Paolozzi L, Wajdula J, Zang C, Nelson H, Raible D. Efficacy and safety of etanercept in moderate-to-severe asthma: a randomised, controlled trial. Eur Respir J. 2011 Jun;37(6):1352-9. doi: 10.1183/09031936.00063510. Epub 2010 Nov 25. PMID 21109557